CLINICAL TRIAL: NCT04751825
Title: Internet-based Emotional Awareness and Expression Therapy for Somatic Symptom Disorder - A Randomized Controlled Trial
Acronym: MBS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm University (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Robert Johansson, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIMBS2
Record Dates: First submitted 2021-02-01; First posted 2021-02-12 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Somatic Symptom Disorder
Keywords: Emotional Awareness and Expression Therapy; Somatic symptom disorder; Central sensitisation; Fibromyalgia; Pain; Self-help; Emotional processing; Trauma
MeSH Terms: conditions — Fibromyalgia; Pain; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: RCT with Wait-List condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-EAET (Experimental): Internet administrated Emotional and Awareness and Expression Therapy (I-EAET). 10 weeks. Self-help treatment with therapist contact via text messages at least once a week.
  Interventions: Behavioral: I-EAET
- WL (No Intervention): Wait-list.

INTERVENTIONS:
Behavioral: I-EAET — See information in arm description.
  Arms: I-EAET

SUMMARY:
The main purpose of this study is to conduct a Randomised Controlled Trial (RCT) where we evaluate an internet administrated version of Emotional Awareness and Expression Therapy (I-EAET) in the treatment of Somatic Symptom Disorder (SSD). We will include 160 patients with SSD that will be randomized to taking part of the Internet based treatment for ten weeks (80 patients) or a waiting list control condition (80 patients). A between-subject design will be used. Self-report measures of symptom level and mechanisms of change will be conducted weekly for the primary outcome measures (PHQ-15, BPI-4) and the process measure (EPS-25). The other self-report measures will be conducted before, after treatment and at follow up at 4-month and 12.

DETAILED DESCRIPTION:
Research background Somatic Symptom Disorder (SSD; DSM-5) is one of the most prevalent disorders encountered in primary care settings (1). Typically in SSD, distressing somatic complaints are accompanied by abnormal thoughts, feelings, and behaviors, emphasizing the role of psychological factors. The experience of somatic symptoms is commonly associated with high levels of impairment in quality of life, psychological distress or increased healthcare utilization (2). In addition, SSD has been associated with an elevated risk for chronic manifestation and comorbid mental disorders, work loss or early retirement (3). Although cognitive behavior therapy (CBT) is the best evidenced psychological treatment for SSD, effect sizes are rather moderate or even small (4). Therefore the question of how to develop more effective treatment protocols for SSD arises.

Difficulties in emotional processing and expression have been demonstrated with patients with SSD in several studies (5). Importantly though, there are indications that an emotion focus in treatment increases the possibility of symptom reduction for patients with SSD (6). In addition, many patients with SSD have experienced stressful/traumatic life events (7). Hence, another potential reason for the limited effect of CBT for SSD may be that these traumas have not been adequately addressed in treatment.

Emotional Awareness and Expression Therapy (EAET) is an affect-focused psychodynamic form of psychotherapy, that has an explicit focus on emotional processing and resolving attachment trauma (8). There is a promising research support for EAET for treating SSD related disorders, where it has been shown to be more effective than CBT in two randomized controlled trials where fibromyalgia and chronic musculoskeletal pain were targeted, respectively (9,10).

Many of today's models of psychotherapy has been tested as guided self-help via the Internet (11). This is a cost-effective, scalable form of psychotherapy delivery. While there exists promising evidence that Internet-based affect-focused psychodynamic therapy is effective in the treatment of depression and anxiety disorders (12,13), there are no published studies on EAET in the format of guided self-help delivered via the Internet.

Preliminary results from a pilot study on Internet-based EAET However, our own group very recently completed a (yet unpublished) pilot trial of Internet based EAET (I-EAET), with an explicit focus on emotional processing using expressive writing. The project was approved by the Swedish Ethical Review Authority (Dnr 2019-03317). We included 52 patients with SSD who took part of a nine-week program based on EAET. Details of the I-EAET intervention are described in the Methods sections below. A large within-group reduction in somatic symptoms (PHQ-15) was observed (Cohen's d = 1.12; 95% CI: 0.77-1.46). Small to moderate magnitude reductions in anxiety (GAD-7), depression (PHQ-9), trauma related symptoms (PCL-5), and dysfunctional emotional processing (EPS25) occurred. Almost one-quarter of the sample (23.1%) achieved a 50% or greater reduction in somatic symptoms. The treatment also significantly increased patient's ability to take part in social and family life (Sheehan Disability Scale). The results were maintained at a four month follow-up. While the results are to be interpreted carefully, the effects seem promising. Further research studies on I-EAET using randomized controlled trials are warranted.

This research proposal is about testing the effects of I-EAET in the treatment of SSD, compared to a waiting-list control condition, using a randomized controlled trial. The long term goal is to develop an intervention that can increase treatment optimization in SSD.

Research questions

a) Can Internet-delivered EAET with an explicit focus on expressive writing decrease bodily symptoms and pain, depression, anxiety and insomnia symptoms, among patients with SSD, as compared to a control condition? b) Is symptom reduction throughout treatment of SSD associated with an increase in emotional processing? c) Are the effects maintained at a 4-month- and 12-month follow-up?

Methods The I-EAET intervention was developed as part of the pilot trial, conducted during late 2019. It is primarily based on Howard Schubiner's book "Unlearn your pain" (14). The I-EAET intervention includes 1) a psychoeducational component on the brain and the nervous system, 2) self-compassion training using meditation techniques, 3) awareness practice on the relationship between trauma, emotions and bodily symptoms, 4) emotional processing using expressive writing exercises, and 5) adaptive interpersonal communication in situations that might trigger pain symptoms. The treatment will last 10 weeks. A secure web-platform (the KI e-Health Core Facility) will be used to provide the treatment via the Internet. Every week the participant in the treatment reads a text consisting of 10-20 pages. The text specifies the theme for the week (i.e. self-compassion) and the home-work assignments to be conducted during the week. Typically, the participants do a daily meditation exercise for 10-15 minutes and an expressive writing assignment for 15-30 minutes. In the daily meditation exercises the participant learn to observe self-critical thoughts and to notice that these thoughts sometimes is anger turned at oneself. Using these meditation exercises, the participants learns to develop a compassionate voice instead of their self-critical one. In the written assignments, usually a stressful or traumatic life event is targeted where emotions are processed in a prespecified order. Emotions tied to these situations are often anger, guilt about anger, sadness and love.

When the participants have done the homework for the week, they send it to their designated psychologist and get written feedback.

Randomized controlled trial of Internet-based EAET for SSD The main purpose of this study is to conduct a Randomised Controlled Trial (RCT) where we evaluate an internet administrated version of Emotional Awareness and Expression Therapy (I-EAET) in the treatment of Somatic Symptom Disorder (SSD). We will include 160 patients with SSD that will be randomized to taking part of the Internet based treatment for ten weeks (80 patients) or a waiting list control condition (80 patients). A between-subject design will be used. Self-report measures of symptom level and mechanisms of change will be conducted weekly for the primary outcome measures (PHQ-15, BPI-4) and the process measure (EPS-25). The other self-report measures will be conducted before, after treatment and at follow up at 4-month and 12.

Feedback on content, process and potential caveats will be collected using surveys and written evaluations from the participants at post-treatment. Linear mixed models will be used to investigate trajectories of change in symptoms and processes.

Time plan January 2021: Recruitment, screening procedure and diagnostic interviews February 2021: Treatment start + Pre-treatment measures conducted April 2021: Treatment ends + Post-treatment measures conducted September 2021: Four-month follow-up + Treatment offered to patients on waiting-list April 2022: Twelve-month follow-up measures

Significance An EAET intervention conducted through the Internet, with a strong focus on emotional processing using expressive writing could potentially increase treatment optimization in SSD and offer a new potential treatment avenue. Furthermore, although several theoretical models of SSD exist, the field lacks solid empirical results from treatment trials, where the analyses of mechanisms of change are conducted using state-of-the-art methods. Such analyses could help to pinpoint the relation between symptom change and emotional processing throughout different phases of treatment.

Ethical considerations Given that the treatment manual in our studies has not been evaluated before, special considerations will be given to adverse effects. As weekly symptom measures will be conducted, we will be able to monitor patients closely for any potential deterioration that will need to be handled. Medical experts will be available for consultation throughout the treatment periods. Adverse events of treatment will also be monitored by using the Negative Effects Questionnaire (NEQ).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* A total score ≥5 on the PHQ-15
* A diagnosis of SSD according to the DSM-5, i.e ≥1 of the 3 of: disproportionate thoughts about the somatic symptom, persistently high level of anxiety, or excessive time and energy devoted in regard to symptoms or health concerns
* Symptom duration ≥6 months
* Written statement from a medical professional that states that a medical evaluation has been conducted.

Exclusion Criteria:

* Alcohol or substance addiction
* A diagnosis of a psychological condition that might require other treatment (e.g., psychosis, suicidality, etc)
* Other severe medical condition
* Ongoing psychological intervention or psychotherapy that target somatic symptoms
* Ongoing medical treatment that may interfere with the psychological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-15. Min (0), Max (30), higher score indicate more somatic symptoms | Baseline
  Measuring somatic symptoms
Patient Health Questionnaire-15. Min (0), Max (30), higher score indicate more somatic symptoms | Post-intervention (10 weeks from start)
  Measuring somatic symptoms
Patient Health Questionnaire-15. Min (0), Max (30), higher score indicate more somatic symptoms | FU at 4 months
  Measuring somatic symptoms
Patient Health Questionnaire-15. Min (0), Max (30), higher score indicate more somatic symptoms | FU at 12 months
  Measuring somatic symptoms
Brief Pain Inventory -4, min (0), max (40) higher score indicate more severe symptoms | Baseline
  Measuring pain symptoms
Brief Pain Inventory -4, min (0), max (40) higher score indicate more severe symptoms | Post-intervention (10 weeks from start)
  Measuring pain symptoms
Brief Pain Inventory -4, min (0), max (40) higher score indicate more severe symptoms | FU at 4 months.
  Measuring pain symptoms
Brief Pain Inventory -4, min (0), max (40) higher score indicate more severe symptoms | FU at 12 months.
  Measuring pain symptoms

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7, min (0), max (21), higher score indicate more severe symptoms | Baseline
  Measuring anxiety symptoms
Generalized Anxiety Disorder-7, min (0), max (21), higher score indicate more severe symptoms | Post-intervention (10 weeks from start)
  Measuring anxiety symptoms
Generalized Anxiety Disorder-7, min (0), max (21), higher score indicate more severe symptoms | FU at 4 month
  Measuring anxiety symptoms
Generalized Anxiety Disorder-7, min (0), max (21), higher score indicate more severe symptoms | FU at 12 month
  Measuring anxiety symptoms
Patient Health Questionnaire-9, min (0), max (27), higher score indicate more severe symptoms | Baseline
  Measuring depressive symptoms
Patient Health Questionnaire-9, min (0), max (27), higher score indicate more severe symptoms | Post-intervention (10 weeks from start)
  Measuring depressive symptoms
Patient Health Questionnaire-9, min (0), max (27), higher score indicate more severe symptoms | FU at 4 month
  Measuring depressive symptoms
Patient Health Questionnaire-9, min (0), max (27), higher score indicate more severe symptoms | FU at 12 month
  Measuring depressive symptoms
Post-traumatic Stress Disorder CheckList-5, min (0), max (80), higher score indicate more severe symptoms | Baseline
  Measuring post traumatic symptoms
Post-traumatic Stress Disorder CheckList-5, min (0), max (80), higher score indicate more severe symptoms | Post-intervention (10 weeks from start)
  Measuring post traumatic symptoms
Post-traumatic Stress Disorder CheckList-5, min (0), max (80), higher score indicate more severe symptoms | FU at 4 month
  Measuring post traumatic symptoms
Post-traumatic Stress Disorder CheckList-5, min (0), max (80), higher score indicate more severe symptoms | FU at 12 month
  Measuring post traumatic symptoms
Shehan Disability Scale (SDS), min (0), max (30), higher score indicate more severe disability | Baseline
  Measuring activity level in three domains (social, work and leisure time)
Shehan Disability Scale (SDS), min (0), max (30), higher score indicate more severe disability | Post-intervention (10 weeks from start)
  Measuring activity level in three domains (social, work and leisure time)
Shehan Disability Scale (SDS), min (0), max (30), higher score indicate more severe disability | FU at 4 month
  Measuring activity level in three domains (social, work and leisure time)
Shehan Disability Scale (SDS), min (0), max (30), higher score indicate more severe disability | FU at 12 month
  Measuring activity level in three domains (social, work and leisure time)
Epworth Sleepiness Scale, min (0), max (24) higher score indicate more severe symptoms | Baseline
  Measuring sleepiness symptoms from
Epworth Sleepiness Scale, min (0), max (24) higher score indicate more severe symptoms | Post-intervention (10 weeks from start)
  Measuring sleepiness symptoms from
Epworth Sleepiness Scale, min (0), max (24) higher score indicate more severe symptoms | FU at 4 month
  Measuring sleepiness symptoms from
Epworth Sleepiness Scale, min (0), max (24) higher score indicate more severe symptoms | FU at 12 month
  Measuring sleepiness symptoms from
Insomnia Severy Index, min (0), max (21), higher score indicate more severe symptoms | Baseline
  Measuring insomnia symptoms
Insomnia Severy Index, min (0), max (21), higher score indicate more severe symptoms | Post-intervention (10 weeks from start)
  Measuring insomnia symptoms
Insomnia Severy Index, min (0), max (21), higher score indicate more severe symptoms | FU at 4 month
  Measuring insomnia symptoms
Insomnia Severy Index, min (0), max (21), higher score indicate more severe symptoms | FU at 12 month
  Measuring insomnia symptoms
Negative Effects Questionnaire, min (0), max (128), higher score indicate more severe negative effects | Post-intervention (10 weeks from start)
  Measuring Negative Effects
Negative Effects Questionnaire, min (0), max (128), higher score indicate more severe negative effects | FU at 12 months
  Measuring Negative Effects
Level of Emotional Awareness Scale, min (0), max (100), higher score indicate better emotional awareness capacity | Baseline
  Measuring emotional awareness capacity
Level of Emotional Awareness Scale, min (0), max (100), higher score indicate better emotional awareness capacity | FU 4 month
  Measuring emotional awareness capacity
Emotional Processing Scale-25, min (0), max (225), higher score indicates more pronounced difficulties with emotional processing capacity | Baseline
  Measuring emotional processing capacity
Emotional Processing Scale-25, min (0), max (225), higher score indicates more pronounced difficulties with emotional processing capacity | Post-intervention (10 weeks from start)
  Measuring emotional processing capacity
Emotional Processing Scale-25, min (0), max (225), higher score indicates more pronounced difficulties with emotional processing capacity | FU 4 month
  Measuring emotional processing capacity
Emotional Processing Scale-25, min (0), max (225), higher score indicates more pronounced difficulties with emotional processing capacity | FU at 12 months
  Measuring emotional processing capacity

OTHER OUTCOMES:
Process measure: Generalized Anxiety Disorder-2, min (0), max (6), higher score indicates more pronounced symptoms | During treatment: Once every week for 10 weeks
  Measuring anxiety symptoms
Process measure: Patient Health Questionnaire-2, min (0), max (6), higher score indicates more pronounced symptoms | During treatment: Once every week for 10 weeks
  Measuring depressive symptoms
Process measure: Emotional Processing Scale-25, min (0), max (225), higher score indicates more pronounced difficulties with emotional processing capacity | During treatment: Once every week for 10 weeks
  Measuring emotional processing capacity
Process measure: Patient Health Questionnaire-15. Min (0), Max (30), higher score indicate more somatic symptoms | During treatment: Once every week for 10 weeks
  Measuring diverse somatic symptoms
Process measure: Brief Pain Inventory-4, min (0), max (40) higher score indicate more severe symptoms | During treatment: Once every week for 10 weeks
  Measuring pain symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Robert Johansson, PhD, Principal Investigator — Karolinska Insitutet
Locations (1):
- Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Background] Budtz-Lilly A, Vestergaard M, Fink P, Carlsen AH, Rosendal M. The prognosis of bodily distress syndrome: a cohort study in primary care. Gen Hosp Psychiatry. 2015 Nov-Dec;37(6):560-6. doi: 10.1016/j.genhosppsych.2015.08.002. Epub 2015 Aug 20. PMID 26371705
- [Background] den Boeft M, Twisk JW, Terluin B, Penninx BW, van Marwijk HW, Numans ME, van der Wouden JC, van der Horst HE. The association between medically unexplained physical symptoms and health care use over two years and the influence of depressive and anxiety disorders and personality traits: a longitudinal study. BMC Health Serv Res. 2016 Mar 22;16:100. doi: 10.1186/s12913-016-1332-7. PMID 27125311
- [Background] Rask MT, Rosendal M, Fenger-Gron M, Bro F, Ornbol E, Fink P. Sick leave and work disability in primary care patients with recent-onset multiple medically unexplained symptoms and persistent somatoform disorders: a 10-year follow-up of the FIP study. Gen Hosp Psychiatry. 2015 Jan-Feb;37(1):53-9. doi: 10.1016/j.genhosppsych.2014.10.007. Epub 2014 Oct 22. PMID 25456975
- [Background] van Dessel N, den Boeft M, van der Wouden JC, Kleinstauber M, Leone SS, Terluin B, Numans ME, van der Horst HE, van Marwijk H. Non-pharmacological interventions for somatoform disorders and medically unexplained physical symptoms (MUPS) in adults. Cochrane Database Syst Rev. 2014 Nov 1;2014(11):CD011142. doi: 10.1002/14651858.CD011142.pub2. PMID 25362239
- [Background] Beck T, Breuss M, Kumnig M, Schussler G. The first step is the hardest - emotion recognition in patients with somatoform disorders. Z Psychosom Med Psychother. 2013;59(4):385-90. doi: 10.13109/zptm.2013.59.4.385. PMID 24307338
- [Background] Farnam A, Somi MH, Farhang S, Mahdavi N, Ali Besharat M. The therapeutic effect of adding emotional awareness training to standard medical treatment for irritable bowel syndrome: a randomized clinical trial. J Psychiatr Pract. 2014 Jan;20(1):3-11. doi: 10.1097/01.pra.0000442934.38704.3a. PMID 24419306
- [Background] Coppens E, Van Wambeke P, Morlion B, Weltens N, Giao Ly H, Tack J, Luyten P, Van Oudenhove L. Prevalence and impact of childhood adversities and post-traumatic stress disorder in women with fibromyalgia and chronic widespread pain. Eur J Pain. 2017 Oct;21(9):1582-1590. doi: 10.1002/ejp.1059. Epub 2017 May 24. PMID 28543929
- [Background] Lumley MA, Schubiner H. Emotional Awareness and Expression Therapy for Chronic Pain: Rationale, Principles and Techniques, Evidence, and Critical Review. Curr Rheumatol Rep. 2019 May 23;21(7):30. doi: 10.1007/s11926-019-0829-6. PMID 31123837
- [Background] Yarns BC, Lumley MA, Cassidy JT, Steers WN, Osato S, Schubiner H, Sultzer DL. Emotional Awareness and Expression Therapy Achieves Greater Pain Reduction than Cognitive Behavioral Therapy in Older Adults with Chronic Musculoskeletal Pain: A Preliminary Randomized Comparison Trial. Pain Med. 2020 Nov 1;21(11):2811-2822. doi: 10.1093/pm/pnaa145. PMID 32451528
- [Background] Lumley MA, Schubiner H, Lockhart NA, Kidwell KM, Harte SE, Clauw DJ, Williams DA. Emotional awareness and expression therapy, cognitive behavioral therapy, and education for fibromyalgia: a cluster-randomized controlled trial. Pain. 2017 Dec;158(12):2354-2363. doi: 10.1097/j.pain.0000000000001036. PMID 28796118
- [Background] Andersson G. Internet-Delivered Psychological Treatments. Annu Rev Clin Psychol. 2016;12:157-79. doi: 10.1146/annurev-clinpsy-021815-093006. Epub 2015 Dec 11. PMID 26652054
- [Background] Johansson R, Bjorklund M, Hornborg C, Karlsson S, Hesser H, Ljotsson B, Rousseau A, Frederick RJ, Andersson G. Affect-focused psychodynamic psychotherapy for depression and anxiety through the Internet: a randomized controlled trial. PeerJ. 2013 Jul 9;1:e102. doi: 10.7717/peerj.102. Print 2013. PMID 23862104
- [Background] Johansson R, Hesslow T, Ljotsson B, Jansson A, Jonsson L, Fardig S, Karlsson J, Hesser H, Frederick RJ, Lilliengren P, Carlbring P, Andersson G. Internet-based affect-focused psychodynamic therapy for social anxiety disorder: A randomized controlled trial with 2-year follow-up. Psychotherapy (Chic). 2017 Dec;54(4):351-360. doi: 10.1037/pst0000147. PMID 29251954
- [Background] Schubiner H, Betzold M. Unlearn your pain : a 28-day process to reprogram your brain. Pleasant Ridge, MI: Mind Body Publishing; 2012.
- [Derived] Maroti D, Lumley MA, Schubiner H, Lilliengren P, Bileviciute-Ljungar I, Ljotsson B, Johansson R. Internet-based emotional awareness and expression therapy for somatic symptom disorder: A randomized controlled trial. J Psychosom Res. 2022 Dec;163:111068. doi: 10.1016/j.jpsychores.2022.111068. Epub 2022 Oct 22. PMID 36327532